CLINICAL TRIAL: NCT05778292
Title: Effect of Different VV ECMO Flows on Lung Perfusion Monitored by EIT: an Observational Study
Brief Title: Effect of Different VV ECMO Flows on Lung Perfusion Monitored by EIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaobo Yang, MD, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: ECMO20221119
Record Dates: First submitted 2023-02-08; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Critical Illness
Keywords: VV ECMO; EIT; Lung perfusion
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate the feasibility of using electric impedance tomography (EIT) to monitor lung perfusion during veno-venous (VV) extracopreal membrane oxygenation (ECMO) support, as well as the effect of different ECMO flows on lung perfusion monitored by EIT.

DETAILED DESCRIPTION:
This is a monocentric obsevensional study that uses EIT to monitor lung perfusion during VV ECMO support and the effect of different ECMO flows on lung perfusion as measured by EIT. Patients on VV ECMO who meet the withdrawal criteria as determined by clinical experts will have their ECMO flow gradually reduced. EIT lung ventilation and perfusion monitoring were performed at various ECMO flows.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 and ≤ 70 years；
2. Patients supported with VV ECMO for respiratory failure；
3. Patients are intubated and mechanically ventilated.

Exclusion Criteria:

1. EIT contraindications such as chest wound dressing, pacemaker installation, defibrillator, etc;
2. Patients who did not sign the informed consent form;
3. Pulmonary embolism;
4. Pneumothorax;
5. Medium to plenty of chest water;
6. Atrial fibrillation or other malignant arrhythmia leads to a decrease in cardiac output;
7. Refractory shock;
8. Severe chronic heart and lung disease has existed in the past;
9. BMI>35 kg/m2;
10. Intra-abdominal pressure >20mmHg.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with respiratory failure supported on VV ECMO
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Lung perfusion at different VV ECMO flows | up to 24hour
  Effect of Different VV ECMO Flows (ECMO flow at 4.5L,3.5L,2.5L,1.5L, and after ECMO withdrawal) on lung perfusion distribution Monitored by EIT

SECONDARY OUTCOMES:
Lung ventilation at different VV ECMO flows | up to 24hour
  Effect of Different VV ECMO Flows (ECMO flow at 4.5L,3.5L,2.5L,1.5L, and after ECMO withdrawal) on lung ventilation distribution monitored by EIT
Lung deadspace region at different VV ECMO flows | up to 24hour
  Effect of Different VV ECMO Flows (ECMO flow at 4.5L,3.5L,2.5L,1.5L, and after ECMO withdrawal) on lung deadspace region monitored by EIT
Lung shunt region at different VV ECMO flows | up to 24hour
  Effect of Different VV ECMO Flows (ECMO flow at 4.5L,3.5L,2.5L,1.5L, and after ECMO withdrawal) on lung shunt region monitored by EIT
Lung ventilation/perfusion matching at different VV ECMO flows | up to 24hour
  Effect of Different VV ECMO Flows (ECMO flow at 4.5L,3.5L,2.5L,1.5L, and after ECMO withdrawal) on lung ventilation/perfusion matching monitored by EIT
Recirculation at different VV ECMO flows | up to 24hour
  Recirculation at different VV ECMO flows (ECMO flow at 4.5L,3.5L,2.5L,and1.5L)

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaobo Yang, Wuhan, Hubei, China